CLINICAL TRIAL: NCT01978457
Title: Establishing and Eliminating Cue-drug Associations in Human Cocaine Addiction
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Not funded
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Robert Malison, Principal Investigator, Yale University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1104008404
Record Dates: First submitted 2013-10-17; First posted 2013-11-07 (Estimated); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Cocaine Dependent Subjects
MeSH Terms: interventions — Cocaine; Propranolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- cocaine hydrochloride (Experimental): cocaine hydrochloride
  Interventions: Drug: cocaine hydrochloride; Drug: propranolol; Drug: placebo
- propranolol (Experimental): propranolol
  Interventions: Drug: cocaine hydrochloride; Drug: propranolol
- placebo (Placebo Comparator): placebo
  Interventions: Drug: cocaine hydrochloride; Drug: propranolol

INTERVENTIONS:
Drug: cocaine hydrochloride
Drug: propranolol
Drug: placebo
  Arms: cocaine hydrochloride

SUMMARY:
We will develop a procedure for conditioning cue-cocaine associations in human drug users. Next, we will reactivate that learning and intervene pharmacologically to prevent the reconsolidation of cue-drug memories. We hypothesize that a combined behavioral and pharmacological approach will have significant potential for persistently inhibiting relapse.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 50 years
2. voluntary, written, informed consent
3. physically healthy by medical history, physical, neurological, ECG, and laboratory examinations
4. DSM-IV criteria for Cocaine Abuse (305.60) or Cocaine Dependence (304.20)
5. recent street cocaine use in excess of that administered in the current study
6. intravenous and/or smoked (crack/freebase) use
7. positive urine toxicology screen for cocaine
8. for females, non-lactating, no longer of child-bearing potential (or agree to practice effective contraception during the study), and a negative serum pregnancy (-HCG) test
9. able to read English and complete study evaluations.

Exclusion Criteria:

1. Other drug dependence (except nicotine)
2. a primary major DSM-IV psychiatric diagnosis (schizophrenia, bipolar disorder, etc.), unrelated to cocaine
3. a history of significant medical (cardiovascular) or neurological illness (e.g., prior myocardial infarction, current active symptoms of cardiovascular disease / angina, evidence of cocaine-related cardiovascular symptoms, prior arrythmias of clinical significance, and/or need for cardiovascular resuscitation, neurovascular events such as transient ischemic attacks, stroke, and/or seizures)
4. current use of psychotropic and/or potentially psychoactive prescription medication
5. seeking treatment for drug abuse/dependence
6. those having contraindications to beta-blocker administration, including diagnoses of asthma, bronchitis, emphysema, or a history of adverse reactions to beta-blockers (including propranolol), as well as those with bradycardia and/or first-degree or greater heart block by ECG

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2012-10; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Total number of patient controlled analgesic (PCA) pump activations (responses) | 3 days
  Data on cocaine self-administration (total number of responses) will be checked for normality prior to analysis using Kolmogorov-Smirnov statistics and normal probability plots. Data that is not normally distributed will be log transformed. If it remains highly skewed after transformation, it will be analyzed using non-parametric approaches (e.g., a non-parametric, ANOVA-Type Statistic). Normally distributed data will be analyzed employing a mixed model design, 3-way ANOVA with co-factors of placebo vs propranolol (between subjects), non-cocaine predicting cues vs. cocaine predicting cues (within subjects) and non-reactivated cocaine cues vs. reactivated cocaine cues (within subjects).

CONTACTS AND LOCATIONS:
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States